CLINICAL TRIAL: NCT04535713
Title: GALLANT: A Phase 2 Study Using Metronomic Gemcitabine, Doxorubicin, Docetaxel and Nivolumab as Second/Third Line Therapy for Advanced Sarcoma
Brief Title: GALLANT: Metronomic Gemcitabine, Doxorubicin, Docetaxel and Nivolumab for Advanced Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-2082
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Doxorubicin; Docetaxel; Nivolumab

STUDY DESIGN:
Intervention Model Description: A total of 260 patients will receive gemcitabine 600 mg/m2 (maximum dose: 1000 mg) on D1 and D8, doxorubicin 18 mg/m2 on D1 and D8 (maximum dose: 32 mg), docetaxel 25 mg/m2 on D1 and D8 (maximum dose: 42 mg), on Days 1 and 8. After the first cycle, nivolumab 240 mg IV will be added on Day 1 of each cycle (see product information; www.accessdata.fda.gov). Treatment cycles are given every 3 weeks. Patients in this study may continue treatment until significant disease progression or unacceptable toxicity occurs up to one year of therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): A total of 260 patients will receive gemcitabine 600 mg/m2 (maximum dose: 1000 mg) on D1 and D8, doxorubicin 18 mg/m2 on D1 and D8 (maximum dose: 32 mg), docetaxel 25 mg/m2 on D1 and D8 (maximum dose: 42 mg), on Days 1 and 8. After the first cycle, nivolumab 240 mg IV will be added on Day 1 of each cycle (see product information; www.accessdata.fda.gov). Treatment cycles are given every 3 weeks. Patients in this study may continue treatment until significant disease progression or unacceptable toxicity occurs up to one year of therapy. Patients who withdraw or do not complete the first 2 treatment cycles and first follow up CT scan/MRI will be replaced.
  Interventions: Drug: Gemcitabine; Drug: Doxorubicin; Drug: Docetaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: Gemcitabine — 600 mg/m2 (Maximum Dose: 1000 mg) i.v. on Day 1 and Day 8 of Cycle 1+
  Other Names: Gemzar
Drug: Doxorubicin — 18 mg/m2 (Maximum Dose: 32 mg) i.v. on Day 1 and Day 8 of Cycle 1+
  Other Names: Adriamycin
Drug: Docetaxel — 25 mg/m2 (Maximum Dose: 42 mg) i.v. on Day 1 and Day 8 of Cycle 1+
  Other Names: Taxotere
Drug: Nivolumab — 240 mg i.v. on Day 1 beginnning Cycle 2+
  Other Names: Opdivo

SUMMARY:
This is an open label phase 2 study for advanced sarcoma using metronomic doses of gemcitabine, doxorubicin and docetaxel, and nivolumab immunotherapy given intravenously.

DETAILED DESCRIPTION:
This is an open label phase 2 study for advanced sarcoma using metronomic doses of gemcitabine, doxorubicin and docetaxel, and nivolumab immunotherapy given intravenously.

A total of 260 patients will receive gemcitabine 600 mg/m2 (maximum dose: 1000 mg) on D1 and D8, doxorubicin 18 mg/m2 on D1 and D8 (maximum dose: 32 mg), docetaxel 25 mg/m2 on D1 and D8 (maximum dose: 42 mg), on Days 1 and 8. After the first cycle, nivolumab 240 mg IV will be added on Day 1 of each cycle (see product information; www.accessdata.fda.gov). Treatment cycles are given every 3 weeks. Patients in this study may continue treatment until significant disease progression or unacceptable toxicity occurs up to one year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of locally advanced, unresectable or metastatic sarcoma
* Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the Investigator's IRB/Ethics Committee
* Willingness to comply with all study procedures and availability for the duration of the study.
* Previously treated patient with measurable disease by RECIST v1.1
* ECOG performance status ≤ 2
* Life expectancy of at least 3 months
* Acceptable cardiac function with LV ejection fraction of > 50%
* Acceptable liver function: Bilirubin < 1.5 times upper limit of normal (ULN; except subjects with Gilbert Syndrome who must have a total bilirubin level < 3.0 ULN); AST (SGOT), ALT (SGPT) and alk phos < 2.5 x ULN (< 5 x ULN if liver metastases present)
* Acceptable renal function: Creatinine < 1.5 times ULN and creatinine clearance > 60 ml/min using the Crockroft-Gault formula
* Acceptable hematologic status: ANC >1000 cells/μL; Platelet count >100,000/μL; Hemoglobin > 9.0 g/dL
* INR and PT < 1.5 ULN unless taking anti-coagulation, in which case PT, INR and aPTT must be within therapeutic range of intended use of anticoagulants
* All women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours of enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; all subjects must agree to use highly effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 5 months for women and 7 months for men after the last dose.

Exclusion Criteria:

* History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Currently receiving treatment with another investigational device or drug study, or <14 days since ending treatment with another investigational device or drug study(s).
* Subject has known sensitivity to gemcitabine, doxorubicin, docetaxel or nivolumab.
* Female subject is pregnant or breast-feeding or planning to become pregnant during study treatment and through 3 months after the last dose of gemcitabine, doxorubicin, docetaxel or nivolumab.
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of gemcitabine, doxorubicin, docetaxel or nivolumab.
* Sexually active subjects and their partners unwilling to use male or female latex condom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  Progression free survival from start of treatment to disease progression or death from any cause

SECONDARY OUTCOMES:
Overall response | 6 weeks
  Overall response by RECIST v1.1 via CT scan or MRI during the treatment period
Adverse Events | 12 months
  Incidence of treatment related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, MD, Principal Investigator — Sarcoma Oncology Research Center, LLC
Locations (1):
- Sant P Chawla, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gordon EM, Sankhala KK, Chawla N, Chawla SP. Trabectedin for Soft Tissue Sarcoma: Current Status and Future Perspectives. Adv Ther. 2016 Jul;33(7):1055-71. doi: 10.1007/s12325-016-0344-3. Epub 2016 May 27. PMID 27234989
- [Result] Demetri GD, von Mehren M, Jones RL, Hensley ML, Schuetze SM, Staddon A, et al. Efficacy and Safety of TRABECTEDIN or Dacarbazine for Metastatic Liposarcoma or Leiomyosarcoma After Failure of Conventional Chemotherapy: Results of a Phase III Randomized Multicenter Clinical Trial. J Clin Oncol. 2015 Sep 14. pii: JCO.2015.62.4734. [Epub ahead of print]. D'Incalci M, Galmarini CM. A Review of TRABECTEDIN (ET-743): A Unique Mechanism of Action. Mol Cancer Ther. 2010; 9:2157-2163.
- [Result] www.accessdata.fda.gov/drugsatfda_docs (Gemcitabine, Doxorubicin, Docetaxel, Nivolumab)
- [Result] Chawla SP, Sankhala KK, Ravicz J, Kang G, Liu S, Stumpf N, Leong B, Kim S, Arasheben S, Tseng WW, Gordon EM. Clinical experience with combination chemo-/immunotherapy using trabectedin and nivolumab for advanced soft tissue sarcoma. J Clin Oncol 36, 2018 (suppl; abstr e23568)
- [Result] Tawbi, HA, Burgess MA, Crowley J et al. Safety and efficacy of PD-1 blockade using pembrolizumab in patients with advanced soft tissue (STS) and bone sarcomas (BS): Results of SARC028-A multicenter phase II study. J Clin Oncol 34, 2016 (suppl; abstr 11006)